CLINICAL TRIAL: NCT03088358
Title: A Multicenter, Randomized, Pilot, Dose-Ranging Clinical Study to Evaluate Safety and Efficacy of TeaRx Xa Factor Direct Inhibitor Versus Enoxaparin as a Venous Thromboembolic Events (VTE) Prevention Following Total Knee Replacement
Brief Title: Safety and Efficacy of TeaRx Xa Factor Direct Inhibitor Versus Enoxaparin as a Venous Thromboembolic Events (VTE) Prevention Following Total Knee Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TeaRx LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CV-TRX-01
Record Dates: First submitted 2017-02-26; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Total Knee Replacement
MeSH Terms: interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TeaRx 50 mg (Experimental): TeaRx: 50 mg per day PO (active 25 mg + placebo 50 mg every 12 hours) during 12 days (±2 days)
  Interventions: Drug: TeaRx
- TeaRx 100 mg (Experimental): TeaRx: 100 mg per day PO (placebo 25 mg + active 50 mg every 12 hours) during 12 days (±2 days)
  Interventions: Drug: TeaRx
- TeaRx 150 mg (Experimental): TeaRx: 150 mg per day PO (active 25 mg + active 50 mg every 12 hours) during 12 days (±2 days)
  Interventions: Drug: TeaRx
- Enoxaparin (Active Comparator): Enoxaparin 40 mg subcutaneous per day (24 hours interval) during 12 days (±2 days)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: TeaRx
  Other Names: TeaRxaban
  Arms: TeaRx 100 mg; TeaRx 150 mg; TeaRx 50 mg
Drug: Enoxaparin
  Other Names: Clexane ®
  Arms: Enoxaparin

SUMMARY:
To evaluate influence of therapy on the following efficacy and safety parameters in different TeaRx dose groups and Enoxaparin group:

* Total venous thromboembolic events (VTE), which includes confirmed deep venous thrombosis (DVT), nonfatal pulmonary embolism (PE), and total mortality
* Incidence of DVT (total, proximal, distal)
* Incidence of nonfatal PE
* Incidence of symptomatic VTE (DVT, PE)
* VTE caused mortality
* Non-VTE caused mortality
* Incidence of all hemorrhagic complications
* Incidence of major and clinically relevant non-major bleeding
* Adverse events (AEs) and serious adverse events (SAEs) from subject complaints, physical examination, vital signs, laboratory results

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years;
* Planned total knee replacement surgery;
* Signed informed consent form;
* Willing to comply with the protocol;
* Willing to use adequate contraception during the trial.

Exclusion Criteria:

* Surgery for acute fracture 4 weeks before screening; history of septic inflammation in the joint; prosthesis revision or one leg missing
* History of venous thrombosis of any location or PE
* History of heparin induced thrombocytopenia or other thrombocytopathy; hemorrhagic diathesis
* History of evident coagulopathy or in a relative
* Congenital thrombophilia
* Bleeding within 6 months of screening; increased risk of bleeding
* BMI less than 18,5 or more than 40 kg/m2
* Systolic BP > 180 mmHg and/or diastolic BP > 110 mmHg registered twice within 15-30 minutes
* Hb ≤ 10.5 g/dL in female or ≤ 11.5 g/dL in male
* Platelets < 100 000/mm3
* Clinical significant abnormalities of APTT and/or INR
* GFR < 30 ml/min/1.73 m2
* ALT or AST ≥ 2 x ULN or total bilirubin ≥1,5 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Incidence of deep venous thrombosis (DVT) (efficacy of the selected TeaRx dose) | 6 weeks following total knee replacement
Incidence of nonfatal pulmonary embolism (PE) (efficacy of the selected TeaRx dose) | 6 weeks following total knee replacement
Incidence of symptomatic venous thromboembolic events (DVT, PE) (efficacy of the selected TeaRx dose) | 6 weeks following total knee replacement
venous thromboembolic events (VTE) caused mortality (efficacy of the selected TeaRx dose) | 6 weeks following total knee replacement
Non-VTE caused mortality (efficacy of the selected TeaRx dose) | 6 weeks following total knee replacement
AEs and SAEs from subject complaints, physical examination, vital signs, laboratory results (efficacy of the selected TeaRx dose) | 6 weeks following total knee replacement

SECONDARY OUTCOMES:
Incidence of bleeding (safety of selected TeaRx dose) | 6 weeks following total knee replacement
  major and clinically relevant non-major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail N. Zamyatin, Prof., Study Chair — Federal State Institution "National Medical and Surgical Center n. a. N. I. Pirogov" of the Ministry of Health of the Russian Federation
Locations (8):
- Russia (8):
  - SHAI "Republican Clinical Hospital of the Ministry of Health of the Republic of Tatarstan", Kazan'
  - Federal State Institution "National Medical and Surgical Center n. a. N. I. Pirogov" of the Ministry of Health of the Russian Federation, Moscow
  - SBEI HPE First Moscow State Medical University n.a. I.M. Sechenov Ministry of Health of the Russian Federation, Moscow
  - SHI of the city of Moscow City Clinical Hospital n.a. S.P. Botkin, Moscow
  - FSBI "Nizhny Novgorod Research Institute of Traumatology and Orthopedics" of the Ministry of Health of the Russian Federation, Nizhny Novgorod
  - SBHI "City Clinical Hospital № 4" of the city of Orenburg, Orenburg
  - St. Petersburg State Institution of Health "City Hospital № 2", Saint Petersburg
  - SHI of the Yaroslavl Region Emergency care hospital n. a. N. V. Solovyov, Yaroslavl

IPD SHARING:
Plan to Share IPD: No